CLINICAL TRIAL: NCT03845764
Title: Interobserver Agreement Between Pulmonologist, Pathologist and Molecular Pathologist in the Assessment of Tumor Burden on ROSE Slides Obtained With Endoscopic Procedures From Pulmonary Nodules and Intrathoracic Lymphadenopathy
Brief Title: Can a Pulmonologist Reliably Assess the Tumor Burden on ROSE Slides Obtained From Pulmonary Nodules and Lymphadenopathy
Status: Completed | Type: Observational
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Principal Investigator, Rocco Trisolini, Director, Interventional Pulmonology Unit, Maggiore Bellaria Hospital, Bologna
Other Study IDs: Bio-Pulmo-ROSE
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rapid on-site evaluation (ROSE): Evaluation, made by a pulmonologist, a pathologist and a molecular pathologist, of the tumor burden in ROSE slides produced from endoscopic procedures aimed at sampling intrathoracic lymphadenopathy and pulmonary nodules
  Interventions: Diagnostic Test: Rapid on-site evaluation

INTERVENTIONS:
Diagnostic Test: Rapid on-site evaluation — Specimens obtained with endoscopic sampling procedures are stained with a rapid method (i.e., Diff Qui) and submitted to on-site cytologic review

SUMMARY:
The study is aimed at verifying if a pulmonologist can reliably assess the tumor burden for the extractive molecular analysis in ROSE samples obtained with endoscopic sampling procedures from intrathoracic lymphadenopathy and pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Indication for endoscopic sampling of suspected malignant lymphadenopathy or pulmonary lesion
* Written informed consent

Exclusion Criteria:

* High risk conditions for the performance of bronchoscopy and/or EBUS-TBNA
* High risk condition for deep sedation (ASA 4)
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with indication to bronchoscopy or endosonography for suspected lung cancer based on imaging (CT and/or PET)
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Accuracy with which a pulmonologist can assess the tumor burden on ROSE slides | The time frame is the duration of each bronchoscopy with endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) for each patient enrolled
  The outcome 1 will be measured by verifying the agreement between the pulmonologist judgment and the molecular pathologist judgment, the latter being the gold standard

SECONDARY OUTCOMES:
Interobserver agreement between pulmonologist, pathologist and molecular pathologist in then assessment of the tumor burden on ROSE slides | The time frame is the duration of each bronchoscopy with endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) for each patient enrolled
  The outcome 2 will be measured by verifying the agreement between the 3 professionals, using the judgment of the molecular pathologist as gold standard
Accuracy with which a pulmonologist can identify malignancy on ROSE samples | The time frame is the duration of each bronchoscopy endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) for each patient enrolled
  The outcome 3 will be measured by verifying the agreement between pulmonologist and pathologist, the latter being the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Policlinico S. Orsola, Bologna
Locations (2):
- Italy (2):
  - Maggiore Hospital, Bologna, Emilia-Romagna
  - Policlinico S. Orsola, Bologna

IPD SHARING:
Plan to Share IPD: No